CLINICAL TRIAL: NCT00332059
Title: Safety and Efficacy Study of Bimatoprost/Timolol Fixed Combination in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-026T
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension | interventions — Bimatoprost

INTERVENTIONS:
Drug: bimatoprost/timolol fixed combination

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Bimatoprost/Timolol Fixed Combination in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of glaucoma or ocular hypertension in both eyes
* Patient requires IOP-lowering drug in both eyes

Exclusion Criteria:

* Uncontrolled medical conditions
* Contraindication to beta-adrenoceptor antagonist therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2003-05; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
IOP

CONTACTS AND LOCATIONS:
Locations (4):
- Bel Air, Maryland, United States
- Vienna, Austria
- Montreal, Quebec, Canada
- Berlin, Germany